CLINICAL TRIAL: NCT00924729
Title: Parallel-group Study of Ocular Penetration of Peri-operative Topically Administered Fluoroquinolones With Cataract Surgery
Brief Title: Study of Ocular Penetration of Topically Administered Fluoroquinolones
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NA_28692
Record Dates: First submitted 2009-06-05; First posted 2009-06-19 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Cataract Extraction
MeSH Terms: interventions — Moxifloxacin; Ophthalmic Solutions; besifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin 0.5% ophthalmic solution (Active Comparator)
  Interventions: Drug: Moxifloxacin 0.5% ophthalmic solution
- Besifloxacin 0.6% ophthalmic suspension (Active Comparator)
  Interventions: Drug: Besifloxacin 0.6% ophthalmic suspension

INTERVENTIONS:
Drug: Moxifloxacin 0.5% ophthalmic solution — Administer moxifloxacin study drug prior to cataract surgery.
  Other Names: Vigamox
  Arms: Moxifloxacin 0.5% ophthalmic solution
Drug: Besifloxacin 0.6% ophthalmic suspension — Administer besifloxacin study drug prior to cataract surgery.
  Other Names: Besivance
  Arms: Besifloxacin 0.6% ophthalmic suspension

SUMMARY:
This study is being conducted to evaluate the intraocular penetration of Moxifloxacin 0.5% ophthalmic solution (Vigamox) and Besifloxacin 0.6% ophthalmic suspension (Besivance) after pre-operative topical administration in subjects undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a visually significant cataract and are planning to have cataract surgery.
* Subjects who are willing/able and have signed informed consent approved by the Institutional Review Board.

Exclusion Criteria:

* Subjects who have a known hypersensitivity, allergy, or contraindication to any fluoroquinolone medication, in any form.
* Subjects who signs of ocular infection or active inflammation in the study eye.
* Subjects who have corneal pathology, including epithelial defect, corneal scarring, or severe dry eye syndrome.
* Subjects who have used any disallowed medication (including antibiotics) during the time period designated as described in the protocol.
* Subjects who have any active or chronic/recurrent ocular or systemic disease that is uncontrolled and is likely to increase the risk of infection to the patient or confound the results of the study.
* Subjects who are pregnant (or suspect to be pregnant) or nursing/lactating.
* Subjects who have participated in any study of an investigational drug or device within 30 days prior to enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Stark, M.D., Principal Investigator — The Wilmer Eye Institute
Locations (1):
- The Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxifloxacin 0.5% Ophthalmic Solution: The patients in this group received one drop of moxifloxacin every 10 minutes for a total of 4 doses, with the last dose given 30+-2 minutes prior to the time of initiating the cataract incision.
- Besifloxacin 0.6% Ophthalmic Suspension: The patients in this group received one drop of besifloxacin every 10 minutes for a total of 4 doses, with the last dose given 30+-2 minutes prior to the time of initiating the cataract incision.
Period: Overall Study
Arm/Group | Moxifloxacin 0.5% Ophthalmic Solution | Besifloxacin 0.6% Ophthalmic Suspension
Started | 25 | 25
Completed | 23 | 25
Not Completed | 2 | 0
Not completed — insufficient volume for analysis | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin 0.5% Ophthalmic Solution | Besifloxacin 0.6% Ophthalmic Suspension | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (8.90) | 68.0 (14.0) | 71.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Aqueous Humor Concentration of Study Drug
Description: Patients were randomly assigned to receive one drop of either moxifloxacin or besifloxacin every 10 minutes for a total of 4 doses, with the last dose given 30 minutes prior to the time of the cataract incision. The aqueous humor was corrected through the paracentesis site. The specimen was transferred immediately to a polypropylene tube and stored upright at ≤ 20° C. Moxifloxacin and besifloxacin concentrations in the aqueous humor were determined using a validated high performance liquid chromatography (HPLC)-tandem mass spectrometry method.
Time Frame: approximately 3 to 4 months
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | Moxifloxacin 0.5% Ophthalmic Solution | Besifloxacin 0.6% Ophthalmic Suspension
Number analyzed (Participants) | 23 | 25
µg/ml | 1.6108 (0.6835) | 0.0312 (0.0131)
Statistical Analysis 1: Comparison: Moxifloxacin 0.5% Ophthalmic Solution vs Besifloxacin 0.6% Ophthalmic Suspension; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Disk Diffusion Assay of Collected Aqueous Humor
Description: A disk diffusion assay was performed to determine the relative antimicrobial activity of the study drug in the aqueous humor. The reference organism used was a clinical isolate of S. epidermidis that will be grown and adjusted to a 0.5 MacFarland turbidity standard. The standardized suspension was inoculated onto a Mueller-Hinton II agar. A sample of the aqueous humor was applied to 6 mm sterile disks, dried, and then placed onto the inoculated Mueller-Hinton II agar plates. The plates were incubated for 24 hours at 35° C. The zone sizes were then recorded.
Time Frame: Approximately 3-4 months.
Population: The amount of aqueous concentration of antibiotic agent was not enough to perform a secondary analysis
Arm/Group | Moxifloxacin 0.5% Ophthalmic Solution | Besifloxacin 0.6% Ophthalmic Suspension
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Moxifloxacin 0.5% Ophthalmic Solution | Besifloxacin 0.6% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes